CLINICAL TRIAL: NCT00685867
Title: An Interventional Study to Evaluate the Impact of Two Innovative Strategies in Preventing Nosocomial MRSA Infection in Surgical Patients
Brief Title: Two Strategies for Methicillin-resistant Staphylococcus Aureus (MRSA) Infection Prevention in Surgical Patients
Acronym: MOSAR-04
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Stephen Harbarth, Professor, University Hospital, Geneva
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LSHP-CT-037940; LSHP-CT-037940
Record Dates: First submitted 2008-05-27; First posted 2008-05-29 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: MRSA Infection
Keywords: Staphylococcus aureus; Resistance; Prevention
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Rapid detection
  Interventions: Other: Rapid molecular MRSA test
- 2 (Other): Enhanced infection control
  Interventions: Behavioral: Hand hygiene promotion

INTERVENTIONS:
Other: Rapid molecular MRSA test — PCR-based rapid screening for MRSA carriage
  Arms: 1
Behavioral: Hand hygiene promotion — * Promotion and monitoring of hand hygiene, with special emphasis on alcohol-based hand rubs and feedback of hand hygiene compliance
  * Standard precautions (e.g. use of gloves for contacts with wounds and body fluids)
  * Isolation precautions according to the hospitals' capacity and strategy
  * Additional basic infection control interventions (if necessary)
  Arms: 2

SUMMARY:
The study is a two-arm controlled multi-centre trial of two strategies to reduce nosocomial MRSA transmission and infection among surgical patients. Enrolment and primary analyses will be performed at the hospital level. A total of ten adult surgical departments with at least 3 surgical subspecialties each will participate in the study. Sites of the study are located in 9 countries (UK, France, Spain, Germany, Switzerland, Italy, Serbia, Greece and Israel).

The primary objective is to determine the effect of an early MRSA detection & decolonization & isolation strategy compared to an enhanced standard control strategy on healthcare-associated MRSA isolation rates among surgical patients at risk of MRSA carriage, who are hospitalized for at least 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Surgical patients with LOS>24h

Exclusion Criteria:

* Surgical patients with LOS<24h

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126750 (Actual)
Dates: Start 2008-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Nosocomial MRSA isolation rate (expressed as the monthly rate of MRSA in clinical isolates divided by the number of susceptible patients per hundred) | Monthly

SECONDARY OUTCOMES:
Nosocomial MRSA infection rate (= number of nosocomial MRSA infections per 100 admissions) | Monthly

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

REFERENCES:
- [Derived] Lee AS, Cooper BS, Malhotra-Kumar S, Chalfine A, Daikos GL, Fankhauser C, Carevic B, Lemmen S, Martinez JA, Masuet-Aumatell C, Pan A, Phillips G, Rubinovitch B, Goossens H, Brun-Buisson C, Harbarth S; MOSAR WP4 Study Group. Comparison of strategies to reduce meticillin-resistant Staphylococcus aureus rates in surgical patients: a controlled multicentre intervention trial. BMJ Open. 2013 Sep 19;3(9):e003126. doi: 10.1136/bmjopen-2013-003126. PMID 24056477